CLINICAL TRIAL: NCT05856669
Title: The Effects of Mirror-Based Virtual Reality Systems and Recalibration Software on Upper Extremity Function in Individuals Experiencing Hemiparesis Post-Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jason Eugene Vice, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300010445
Record Dates: First submitted 2023-04-16; First posted 2023-05-12 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Stroke; Hemiparesis
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single subject case study (Experimental)
  Interventions: Device: Virtual reality gaming

INTERVENTIONS:
Device: Virtual reality gaming — This study aims to combine the motivational delivery of therapy which is an immersive virtual reality with the foundational concepts of mirror therapy. By utilizing a recalibration software, the participant will be able to achieve magnified movements on their screen as compared to the limited movement that is occurring in reality. The recalibration software takes each plane of movement of the gaming controller and magnifies the participant's range of motion in order to promote greater participation and success in the game that they are playing (Walkin VR). By using the fundamental concepts of mirror therapy in an immersive virtual reality setting, the investigators aim to mimic the results of mirror therapy while increasing motivation and adherence to the therapeutic program to increase overall upper extremity function.

SUMMARY:
The goal of this study is to learn about the benefits of using a virtual reality gaming system that can be adjusted for a person who has upper arm weakness from stroke. The main question it aims to answer is whether strength and movement in the upper arm be improved by use of the gaming system.

Participants will be asked to complete initial measurements of upper arm function, play a video game for one hour, four times a week for five weeks, and repeat the measurements of upper arm function at the end.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported diagnosis of stroke
* Greater than 2 years post-stroke
* Access to reliable transportation
* History of weakness/hemiparesis of one upper limb

Exclusion Criteria:

* Significant vision impairment or blindness
* Non-English speaking
* History of seizure or seizure disorder
* Health conditions which would be exacerbated by low-intensity exercise
* Inability to use arms independently for exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Change in upper extremity active range of motion | 6 weeks
  Measured via goniometer
Change in grip strength | 6 weeks
  Measured via hand dynamometer

SECONDARY OUTCOMES:
Change in aerobic fitness | 6 weeks
  Measured via oxygen consumption using a wearable metabolic monitor while pedaling an arm bike

CONTACTS AND LOCATIONS:
Overall Officials: Jason Vice, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Lakeshore Foundation Research Collaborative, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bao X, Mao Y, Lin Q, Qiu Y, Chen S, Li L, Cates RS, Zhou S, Huang D. Mechanism of Kinect-based virtual reality training for motor functional recovery of upper limbs after subacute stroke. Neural Regen Res. 2013 Nov 5;8(31):2904-13. doi: 10.3969/j.issn.1673-5374.2013.31.003. PMID 25206611
- [Result] Mekbib DB, Zhao Z, Wang J, Xu B, Zhang L, Cheng R, Fang S, Shao Y, Yang W, Han J, Jiang H, Zhu J, Ye X, Zhang J, Xu D. Proactive Motor Functional Recovery Following Immersive Virtual Reality-Based Limb Mirroring Therapy in Patients with Subacute Stroke. Neurotherapeutics. 2020 Oct;17(4):1919-1930. doi: 10.1007/s13311-020-00882-x. PMID 32671578
- [Result] Modrono C, Navarrete G, Rodriguez-Hernandez AF, Gonzalez-Mora JL. Activation of the human mirror neuron system during the observation of the manipulation of virtual tools in the absence of a visible effector limb. Neurosci Lett. 2013 Oct 25;555:220-4. doi: 10.1016/j.neulet.2013.09.044. Epub 2013 Sep 27. PMID 24080372